CLINICAL TRIAL: NCT05507099
Title: A Phase 2, Randomized Study to Compare Bone Marrow Aspirate Versus Lipoaspirate Concentrate Autologous Cell Therapy for the Treatment of the Knee and Hip Osteoarthritis in Adults
Brief Title: Stem Cell Study in Osteoarthritis of the Knee and Hip Joints
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grigory Karmy (Other)
Responsible Party: Sponsor-Investigator, Grigory Karmy, Qualified Investigator, Dr. G. Karmy Medicine Professional Corporation
Organization: Dr. G. Karmy Medicine Professional Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Knee arm randomized to Lipoaspirate Concentrate and Bone Marrow Aspirate (Active Comparator): The Subjects will be randomized to one of the treatment groups separately for the knee and hip arms of the study. Group A will receive a single intra-articular injection with lipoaspirate concentrate to the knee and Group B will receive a single intra-articular injection with bone marrow aspirate concentrate.
  Interventions: Biological: Bone Marrow Aspirate, Lipoaspirate Concentrate
- Hip Arm randomized to Lipoaspirate Concentrate and Bone Marrow Aspirate (Active Comparator): The subjects will be randomized to one of the treatment groups separately for the knee and hip arms of the study. Groups C will receive a single intra-articular injection with lipoaspirate concentrate to the hip and Group D will receive a single intra-articular injection with bone marrow aspirate.
  Interventions: Biological: Bone Marrow Aspirate, Lipoaspirate Concentrate

INTERVENTIONS:
Biological: Bone Marrow Aspirate, Lipoaspirate Concentrate — Autologous Cell Therapy.

SUMMARY:
The purpose of this trial is to compare the effect of a single intra-articular injection of Lipoaspirate Concentrate vs Bone Marrow Aspirate on pain reduction and functional improvement in the treatment of the knee and hip OA.

DETAILED DESCRIPTION:
The primary objective is to compare of magnitude and duration of pain relief of intra-articular injections with Lipoaspirate Concentrate vs Bone Marrow Aspirate.

The secondary objective is to compare the effect of Lipoaspirate Concentrate vs Bone Marrow Aspirate intra-articular injections on functional improvement, stiffness, global impression of change, and consumption of analgesic medication.

The exploratory objective is to explore the safety and the general tolerability of a single intra-articular injection of Lipoaspirate Concentrate vs Bone Marrow Aspirate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 95 years old
2. Residents of Canada
3. Written informed consent to participate in the study
4. Willingness and ability to comply with the study procedures and phone visit schedules and ability to follow verbal and written instruction
5. The NRS for at least 5 daily measures will be used to calculate the average score. An average NRS pain score 4-9 (moderate to severe pain).
6. Diagnosis of symptomatic knee or hip osteoarthritis for at least 12 weeks prior to screening based on an X-ray performed within 1 year prior to screening period.
7. Radiographic evidence of OA of the index knee or hip (Kellgren-Lawrence Grade I to IV) within 1 year prior to screening or during the screening period.
8. Failed conservative treatment for more than 12 weeks before the screening, meaning that pain persists for more than 12 weeks after the patient tried two or more of the following medication or interventions in that period.

   * oral analgesics, including over-the-counter medications and supplements,
   * physiotherapy
   * acupuncture
   * bracing
   * cortisone injections,
   * hyaluronic acid injections,
   * dextrose injections (prolotherapy)
   * platelet-rich plasma injections
9. Women of childbearing potential must use an effective method of contraception from 14 days prior to baseline visit to 360 days after intervention. Effective birth control considered for this trial are total abstinence; consistent use of birth control pills; injectable birth control methods; intrauterine device placement; and tubal ligation or male partner with vasectomy; diaphragm with contraceptive jelly or condom with contraceptive foam.This does not apply to male and postmenopausal women.
10. Body mass index (BMI) ≤ 50 kg/m2

Exclusion Criteria:

1. Women who are pregnant or planning to become pregnant during the trial period.
2. Women of childbearing potential (not surgically sterile or post-menopausal for at least one year) not using a highly effective method of contraception such as total abstinence; consistent use of birth control pills; injectable birth control methods; intrauterine device placement; and tubal ligation or male partner with vasectomy; diaphragm with contraceptive jelly or condom with contraceptive foam.
3. History of malignancy except for the diagnosis of basal cell carcinoma, within 5 years prior to pre-screening.
4. Presence of retained rods or screws or insertion or joint replacement in the joint to be injected
5. History of autoimmune diseases including lupus and rheumatoid arthritis
6. Prior arthroscopic or open surgery of the index joint within 6 months prior to screening
7. Planned arthroscopic or open surgery of the index joint during study period
8. Intra-articular injections in the index joint within 3 months prior to screening for corticosteroids or dextrose injections, and within 6 months prior to screening for hyaluronic acid or platelet-rich plasma (PRP) injections
9. Use of systemic immunosuppressives, immunomodulators or chemotherapeutic agents within 3 months prior to baseline visit
10. Know hypersensitivity to lidocaine, epinephrine or heparin
11. History of coagulopathy
12. Fever (forehead temperature above 38.0 centigrade) at baseline visit
13. Subjects with cutaneous infection at the lipoaspirate or bone marrow aspirate site and/or in the area of the injection at baseline visit
14. Subjects with hemoglobin less than 10 g/L
15. Subjects with platelet count less than 155x109/L
16. Subjects participating in a study of an experimental drug or medical device within 30 days of study entry
17. Any medical condition the qualified investigator believes makes the patient unsuitable for the study
18. Subjects using warfarin before the screening, with an INR above 3

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2028-08-08 (Estimated); Study Completion 2028-08-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the change from the Baseline to the Day 360 in WOMAC pain subscale pain subscale | 360 days

SECONDARY OUTCOMES:
Change from Baseline to Days 90, 180 in WOMAC pain subscale | 90, 180 days
Change from Baseline to Days 90, 180, and 360 in WOMAC stiffness subscale | 90, 180, 360 days
Change from Baseline to Days 90, 180, and 360 in WOMAC function subscale | 90, 180, 360 days
Change from Baseline to Days 90, 180, and 360 in total WOMAC score | 90, 180, 360 days
Change from Baseline to Days 90, 180, and 360 in Patient's Global Impression of Changes (PGIC) | 90, 180, 360 days
Change in average weekly consumption of analgesic medications from Baseline to Day 90, 180, and 360 | 90, 180, 360 days

CONTACTS AND LOCATIONS:
Overall Officials: Grigory Karmy, MD, Principal Investigator — McMaster University
Locations (1):
- Karmy Clinic, Brampton, Ontario, Canada